CLINICAL TRIAL: NCT02960945
Title: An Open-Label Single-Dose Crossover Pharmacokinetic Study to Compare CTP-543 to Jakafi® in Healthy Volunteers
Brief Title: Open-Label Crossover Study Comparing CTP-543 to Jakafi®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CP543.1002
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Healthy
MeSH Terms: interventions — Tablets; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CTP-543 (Experimental): Tablet, single oral dose
  Interventions: Drug: CTP-543, 16 mg (2 x 8 mg tablet)
- Jakafi (Active Comparator): Tablet, single oral dose
  Interventions: Drug: Jakafi 15Mg Tablet

INTERVENTIONS:
Drug: CTP-543, 16 mg (2 x 8 mg tablet)
  Arms: CTP-543
Drug: Jakafi 15Mg Tablet
  Arms: Jakafi

SUMMARY:
This study will assess the metabolite and pharmacokinetic (PK) profile of a single dose of CTP-543 compared to a single dose of Jakafi® in healthy volunteers.

DETAILED DESCRIPTION:
The crossover design will assess the safety, tolerability, PK and metabolite profiles of a single dose of CTP-543 compared to a single dose of Jakafi. Approximately 12 healthy volunteers will be enrolled in this open label study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females between 18 and 50 years of age, inclusive
* Body weight ≥ 50 kg and BMI within the range of 18 to 30 kg/m2, inclusive

Exclusion Criteria:

* History of clinically significant central nervous system (eg, seizures), cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal (GI) conditions
* PR interval > 220 msec or QRS duration > 120 msec or QTcF interval > 450 msec obtained at screening visit or prior to the first dose of study drug
* History of herpes zoster
* Hemoglobin, white blood cell, or platelet levels below the lower reference limit at screening or prior to the first dose of study drug
* Liver function tests greater than the upper limit of normal
* Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody
* Urinalysis positive for protein or glucose
* A positive screen for alcohol, drugs of abuse, or tobacco use
* Donation of blood, plasma or other blood products prior to screening
* A positive tuberculosis test

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Measurement of CTP-543 metabolites and exposure in plasma under fasted conditions | 24 hours

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 24 hours
Measurement of CTP-543 metabolites and exposure in urine under fasted conditions | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No